CLINICAL TRIAL: NCT00678470
Title: A Single Arm, Open Label Study to Explore if Response to Intralesional Alefacept Injections Prior to the Standard Course of Intramuscular Treatment Can Predict Clinical Outcomes in Patients With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: Open Label Study of Alefacept Injections to Patients With Moderate to Severe Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Tina Bhutani, Principle Investigator, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KOO-AMEVIVE-2008; CHR-H5939-31199-01 (Other: UCSF Committee for Human Research)
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Results first posted 2013-02-15 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Moderate to Severe Psoriasis
MeSH Terms: interventions — Alefacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): Investigational intervention without random assignment
  Interventions: Drug: Intralesional Alefacept

INTERVENTIONS:
Drug: Intralesional Alefacept — Patients enrolled in this study will receive intralesional alefacept injections to a single psoriatic plaque at week 0. After a two week observation period, patients will receive 15 mg intramuscular alefacept for 12 weeks.
  Other Names: Amevive

SUMMARY:
This is a single-center, open-label, pilot study. A total of 18 subjects will be enrolled in this 6 month study to evaluate whether the response to intralesional alefacept injections prior to the standard course of intramuscularly (IM) treatment can predict clinical outcomes in psoriasis patients. One lesion with a psoriasis severity assessment score greater than 3 and an induration score greater than 1 will be identified on each patient. Each lesion will receive only one intralesional alefacept injection during the first three weeks of the study (1 lesion per week). Following a 2 week observation period, subjects will undergo a standard 12 week course of weekly intramuscular alefacept injections. The Psoriasis Area Severity Index (PASI) score will be used to determine the effectiveness of the intramuscular alefacept treatments. An 8 week follow-up period will begin after the last dose of alefacept is administered where safety and efficacy measures will continue to be monitored as outlined in the study procedures. The hypothesis is that the response to intralesional alefacept injections, whether it is positive or no benefit, will predict the clinical response to intramuscular alefacept administration.

DETAILED DESCRIPTION:
See Brief Summary

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are nonimmunocompromised males or females 18 years of age or older
2. Subjects have moderate to severe plaque-type psoriasis.
3. Subjects have a Body Surface Area (BSA) involvement of greater than 5%.
4. Subjects have a Psoriasis Area and Severity Index (PASI) greater than 10.
5. Subjects have three psoriatic lesions with psoriasis severity score greater than or equal to 6 and an induration score greater than or equal to 2.
6. Subjects' target lesions are greater than 2 cm2 preferably on similar anatomical regions.
7. Subjects are eligible for systemic therapy, particularly alefacept, in the opinion of the investigator.
8. Before any study-specific procedure, subject must sign/date the appropriate written informed consent, HIPAA authorization, and a photography consent form.
9. Negative urine pregnancy test within 7 days before the first dose of alefacept in all women (except those surgically sterile or at least 1 years postmenopausal)
10. Subjects must be in general good health with no other skin disease, state of physical condition which would impair evaluation of psoriasis or which would increase their health risk by study participation.
11. Subject agrees to comply with protocol requirements, attend all regularly study visits and is considered to be a good study subject.
12. Subject meets concomitant medication washout requirements.

Exclusion Criteria:

1. Subjects with erythrodermic, pustular, or guttate psoriasis.
2. Evidence of skin conditions other than psoriasis that would interfere with study-related evaluations of psoriasis.
3. Subject has a known sensitivity to any component of the study medications.
4. Evidence of active infections such as fevers, chills, sweats, or history of untreated Lyme disease and active severe infections within 4 weeks before screening visit, or between the screening and Week 0 visits.
5. Subjects whose CD4+ T-lymphocyte count at study entry is less than the lower limit of normal per reference laboratory.
6. History of immune compromised status [e.g. human immunodeficiency virus (HIV) positive status or other immune suppressing drug] or a congenital or acquired immunodeficiency.
7. Subject has a poorly controlled medical condition including, but not limited to, unstable cardiovascular disease, poorly controlled diabetes, recent stroke, history of recurrent infections, or any other condition for which, in the opinion of the investigator, participation in the study would place the subject at risk.
8. Subject has a history of or ongoing drug or alcohol abuse.
9. Female subjects who are not postmenopausal for at least 1 year, surgically sterile, or willing to practice effective contraception during the study. Nursing mothers, pregnant women and women planning to become pregnant while on study are to be excluded.
10. Subject plans to receive any live vaccines during the study.
11. Current enrollment in another clinical study and treatment with another experimental drug or approved therapy for experimental use within 30 days prior to Week 0.
12. Subjects that cannot commit to all the assessments required by the protocol.
13. Any disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures.
14. Subject is considered by the investigator, for any reason, to be an unsuitable candidate for study participation.
15. Subjects that cannot or do not wish to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Koo, MD, Principal Investigator — UCSF Psoriasis and Skin Treatment Center, Department of Dermatology, University of California, San Francisco
Locations (1):
- UCSF Psoriasis and Skin Treatment Center, San Francisco, California, United States

REFERENCES:
- [Result] Bhutani T, Kamangar F, Zitelli K, Chiang C, Gattu S, Nguyen T, Becker E, Koo J. Intralesional injections of alefacept may predict systemic response to intramuscular alefacept: results from a pilot study. J Dermatolog Treat. 2013 Oct;24(5):348-50. doi: 10.3109/09546634.2012.672712. Epub 2012 Jun 5. PMID 22506829

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from our medical clinic as well as through flyers posted at other University of California at San Francisco sites.
Pre-assignment Details: Patients were required to have a 2 week washout from topicals and one month washout from any systemic agents.
Groups:
- Intralesional Alefacept: Investigational intervention without random assignment
  Intralesional Alefacept : Patients enrolled in this study will receive intralesional alefacept injections once a week for 3 weeks in three different lesions. Each lesion will only be injected once with one alefacept concentration. The week it is administered will depend on the concentration. Three different concentrations of the alefacept preparation will be administered.
Period: Overall Study
Arm/Group | Intralesional Alefacept
Started | 18
Completed | 14
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Intralesional Alefacept
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Either or Both Intralesional Response and Systemic Response
Description: Target plaque assessment completed using local Physician's Global Assessment score (PGA). Systemic response measured by comparing Psoriasis Area and Severity Index score at week 22 compared to baseline. Correlation measured using Fisher's non parametric test of association.
Time Frame: 22 weeks
Population: Eighteen patients were enrolled in the study and 14 patients completed the entire 22-week protocol. Three patients were lost to follow-up. One patient was discontinued due to persistent elevated liver enzymes determined by the investigators as secondary to heavy alcohol use.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 14
Participants
  Systemic Resp:IL Resp | 8
  Systemic Resp:IL Nonresp | 0
  Systemic Nonresp:IL Resp | 0
  Systemic Nonresp:IL Nonresp | 6
Statistical Analysis 1: Comparison: Single Arm; Test type: Other; p = 0.0003, Fisher Exact; Correlation = 1; Using Fisher's non-parametric test of associations, correlations were determined between the patients who were intralesional responders with their response at ‡70% change in PASI score

ADVERSE EVENTS:
Arm/Group | Intralesional Alefacept
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes